CLINICAL TRIAL: NCT06069219
Title: Pharmacokinetics of Sufentanil After Epidural Administration in Patients Undergoing Abdominal Surgery
Brief Title: Pharmacokinetics of Sufentanil After Epidural Administration
Status: Completed | Type: Observational
Sponsor: Poznan University of Medical Sciences (Other)
Collaborators: Medical University of Gdansk (Other); Clinical Hospital Heliodor Swiecicki of the Medical University of Karol Marcinkowski in Poznań (Other)
Responsible Party: Principal Investigator, Agnieszka Bienert, Full Professor, Poznan University of Medical Sciences
Other Study IDs: 1144/18; 2014/15/N/NZ7/03028 (Other Grant/Funding Number: Polish National Science Centre)
Record Dates: First submitted 2023-10-01; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-10

CONDITIONS: Epidural; Anesthesia; Epidural Analgesia; Abdominal Surgery
Keywords: abdominal surgery; epidural analgesia; epidural anesthesia; pharmacokinetics; surgery patients; sufentanil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients received epidural sufentanil during and after abdominal surgery: All patients were premedicated with oral midazolam 7,5 mg and then they were induced into general endotracheal anesthesia according to a standardized protocol, with propofol 1-3 mg/kg, fentanyl 1-2 ug/kg and rocuronium bromide 0.6 mg/kg. Anaesthesia was continued with sevoflurane or desflurane MAC 1 to maintain mean arterial pressure with a value of +/- 20% of the original value. The epidural sufentanil infusion was started with bolus during anesthesia and continued after surgery as long as was necessary.
  Interventions: Drug: Epidural administration of sufentanil

INTERVENTIONS:
Drug: Epidural administration of sufentanil — The epidural cannulations were placed by anesthesiologists before general anesthesia. Correct positioning of the catheters were tested and confirmed by negative aspiration and injection of 3 mL of 2% Lidocaine. The epidural infusion (solution of 0.2 % ropivacaine 5 ml with 25 to 50 mcg sufentanil in 50 ml of 0,9% NaCl) was started with bolus of 5 ml over 5 minutes and then continuous infusion was maintained was throughout the surgery at 3-12 mL/h and 2-12 mL/h after the surgery. Single dose of sufentanil was given when needed.
  Other Names: Continuous epidural infusion of sufentanil

SUMMARY:
Sufentanil is an opioid analgesics used in all groups of patients. It has one of the strongest effects among analgesic drugs. Sufentanil is widely-used because of its very quick onset, short duration of action, and better hemodynamic stability in patients compared to other opioids. Most of the pharmacokinetic studies described intravenous administration of sufentanil. The drug can also be epidural administrated (especially continuous epidural infusion) in low concentration with local anesthetics (ropivacaine or bupivacaine) for epidural analgesia. Epidural analgesia offers effective pain relief not only during the surgery, but also postoperatively. The combination of two drugs provides their additive effect and can reduce doses required for pain relief, then decreases the number and severity of adverse events. The study aims to describe the pharmacokinetics of epidural sufentanil used perioperative in adult patients after abdominal surgery to adjust the dosage if necessary.

DETAILED DESCRIPTION:
The patients qualified for abdominal surgery were enrolled in the study. All patients were premedicated with oral midazolam (7.5 mg). Epidural cannulations were placed by anesthesiologists before general anesthesia. The catheters' placement procedure was conducted under local anesthesia and according to the local protocol for the infections' prevention. The epidural infusion (solution of 0.2 % ropivacaine 5 ml with 25 to 50 mcg sufentanil in 50 ml of 0,9% NaCl) was started with a 5 mL bolus of the mentioned solution a few minutes before skin incision. The continuous infusion was maintained throughout the surgery at the rate of 3-12 mL/h. The patients were induced into general endotracheal anesthesia according to a standardized protocol, with propofol 1-3 mg/kg, fentanyl 1-2 mcg/kg, and rocuronium bromide 0.6 mg/kg. Anaesthesia was continued by using sevoflurane or desflurane MAC 1 to maintain mean arterial pressure with a value of +/- 20% of the original value. The postoperatively patients were monitored in the PACU (Post Anesthesia Care Unit) for 1 hour and then transferred to the intensive care unit or surgical unit according to their clinical status and co-morbidities. Whole blood samples (2.0 ml) were collected to measure sufentanil concentrations - during the epidural infusion and up to 72 hours after its cessation. Vital parameters (e.g. blood pressure, saturation, heart rate, respiratory rate, and pain score) were monitored at regular intervals. The epidural sufentanil and ropivacaine infusion were continued after surgery as long as was necessary.

ELIGIBILITY:
Inclusion Criteria:

* age 18-70 years,
* qualifications for abdominal surgery,
* ASA I-III

Exclusion Criteria:

* proven allergies to sufentanil,
* lack of written confirmed consent of a patient

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The adult patients qualified to abdominal surgery performed in epidural anesthesia using sufentanil.
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Measurement of the depth of analgesia using NRS | before the beginning of sufentanil administration, during sufentatnil administration, up to 72 hours after sufentatnil administration
  Measurement of the depth of analgesia using NRS (Numeral Rating Scale) during epidural administration of sufentanil. Sufentanil was given for surgery patients during and after abdominal surgery as an analgesic agent.
Sufentanil plasma concentrations [pg/ml] | 5, 30 minutes, 1, 2, 4, 6, 12 h after the begining of epidural infusion of sufentanil, then 1 blood samples every 24 h, just before the epidural infusion cessation and 3, 5, 20, 40 minutes, and 1, 2, 6, 12, 36, 72 hours after the infusion cessati
  Measurements of sufentanil plasma concentrations [pg/ml] during epidural analgesia with sufentanil. Whole blood samples (2.0 ml) were collected according to the study protocol.
Systolic blood pressure | before the beginning of sufentanil administration, during sufentatnil administration, up to 72 hours after the cessation of sufentatnil administration
  Measurements of systolic blood pressure during epidural analgesia with sufentanil.
Diastolic blood pressure | before the beginning of sufentanil administration, during sufentatnil administration, up to 72 hours after the cessation of sufentatnil administration
  Measurements of diastolic blood pressure during epidural analgesia with sufentanil.
Heart rate | before the beginning of sufentanil administration, during sufentatnil administration, up to 72 hours after the cessation of sufentatnil administration
  Measurements of heart rate during epidural analgesia with sufentanil.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Grześkowiak, MSc, PhD, Study Director — Poznan University of Medical Sciences; Krzysztof Kusza, MD, PhD, Study Director — Heliodor Swiecicki Clinical Hospital in Poznan
Locations (2):
- Poland (2):
  - Heliodor Swiecicki Clinical Hospital in Poznan, Poznan, Greater Poland Voivodeship
  - Medical University of Gdansk, Gdansk, Pomeranian Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
All data with analysis will be available after a publication of study results as a manuscript.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available in 12 months and available for 5 years
Access Criteria: Scientists

REFERENCES:
- [Derived] Bienert A, Moor AB, Okunska P, Ber J, Siluk D, Waszczuk M, Kusza K, Bartkowiak T, Szrama J, Kluzik A, Koszel T, Wiczling P. Pharmacokinetics of Sufentanil After Epidural Administration During the Course of Extensive Abdominal Surgery. Clin Pharmacokinet. 2025 Sep;64(9):1331-1340. doi: 10.1007/s40262-025-01543-y. Epub 2025 Jun 29. PMID 40581890